CLINICAL TRIAL: NCT04638062
Title: Effect of Post Isometric Relaxation Versus Myofascial Release Therapy on Pain, Functional Disability and QoL in the Management of Non Specific Neck Pain: A Randomized Controlled Trial
Brief Title: Effect of Post Isometric Relaxation Versus Myofascial Release Therapy in the Management of Non Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Zainab Khalid Khan, Physiotherapist, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DUHS/IPMR/000
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Neck Pain
Keywords: Non specific neck pain; Post isometric relaxation; Muscle energy techniques; Myofascial Release therapy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Isometric Relaxation (Experimental): This study ARM will receive following therapies
  1. Post isometric relaxation (Upper Trapezius and Levator Scapulae muscles)
  2. Isometric neck strengthening exercises
  3. Cryotherapy
  Interventions: Other: 1.Post Isometric Relaxation
- Myofascial Release Therapy (Experimental): This study ARM will receive following therapies
  1. Myofascial release therapy (Upper Trapezius and Levator Scapulae muscles
  2. Isometric neck strengthening exercises
  3. Cryotherapy
  Interventions: Other: 1.Myofascial Release therapy

INTERVENTIONS:
Other: 1.Post Isometric Relaxation — For Upper Trapezius In supine position Neck flexion, contra-lateral full side bending followed by slight ipsilateral rotation will be provided towards the side being treated. while asking the patient to shrug the stabilized shoulder and contraction will be maintained for 7- 10s. Repeating it 3-5 times.
  For Levator Scapulae Step One In supine position while lifting the patients neck in full flexion, lateral flexion and rotation with 7-10s isometric contraction away from side to be treated will be provided.
  Step Two The patient will be instructed to take head backwards to the table while at the same time asking the patient to slightly shrug the shoulder and resistance will be provided. Repeating it 3-5 times.
  2.Neck isometric strengthening exercises Intensity 5 reps Frequency at 1st week one set and second week will progress to 2 sets
  3.Cryotherapy will be placed on cervical region for 10 min after the treatment.
  Arms: Post Isometric Relaxation
Other: 1.Myofascial Release therapy — For Upper Trapezius In sitting position Myofascial Release of Trapezius will be performed unilaterally with soft fist or elbow sinking and then taking up the line of tension from mid belly of Trapezius, to the acromion process, while the patient drops the head forward and will slowly rotate the head from side to side. While providing the resistance to contralateral side of rotation. Repeating for 2-3 times.
  For Levator Scapulae In sitting position applying same unilateral muscle release as Trapezius, but the line of tension will be to the inferior border of Scapulae slightly laterally and will ask the patient to drop the head forward to increase resistance on Levator muscle. Repeating it 2-3 times
  2.Neck isometric strengthening exercises Intensity 5 reps Frequency at 1st week one set and second week will progress to 2 sets
  3.Cryotherapy will be placed on cervical region for 10 min after the treatment.
  Arms: Myofascial Release Therapy

SUMMARY:
Non-specific neck pain (NS-NP) is the most prevailing musculoskeletal disorder (MSK) which has large socio-economic burden worldwide. It is associated with poor posture and neck strain which may lead to pain and restricted mobility. Post isometric relaxation a form of Muscle energy technique, that works on the principles of restoring biomechanics, reducing the movement restriction and pain. Myofascial release therapy will improve muscle immobility and pain by improving blood circulation lymphatic drainage and relaxing the contracted muscles. The aim of this study is to determine the effect of Post-isometric relaxation Versus Myofascial release therapy on pain, range of motion, disability and quality of life in the management of non-specific neck pain.

DETAILED DESCRIPTION:
A randomized control trial will be conducted at IPMR (Institute of Physical Medicine and Rehabilitation) on 60 patients with non-specific neck pain with age group between 25-40 years. Initial screening of the patients will be carried out by referring physiatrist. Patients who fulfils inclusion criteria will be randomly allocated to either group by computer generated random sampling after taking written informed consent. All the patients will be evaluated using Visual analogue scale for pain, Neck disability index for functional status and disability, Universal goniometer for cervical range of motion and WHO BREF for quality of life on 1st and 6th sessions. Group 1 will receive Post isometric relaxation for Upper trapezius and levator scapulae along with Cryotherapy and strengthening exercises . Group 2 will receive myofascial release therapy for Upper Trapezius and Levator scapulae muscles along with cryotherapy and strengthening exercises. Data will be analyzed using the SPSS version 21. Baseline reading will be taken for further comparison at the end of treatment. Baseline variables are Pain, ROM, Functional disability and Qol. For within group analysis, paired sample t test will be used. For intergroup independent sample t test will be used. P value less than 0.05 will be set as threshold to detect statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Non-specific neck pain for 2-6 weeks.
2. Unilateral neck pain
3. Patients' age group between 25 - 40.
4. On VAS scale pain intensity >4.

Exclusion Criteria:

1. Cervicogenic headache.
2. Tumor of cervical spine.
3. Whiplash injury.
4. Cervical Fractures
5. Normal ROM of cervical spine.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-11-20 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | baseline and post intervention 2 weeks
  NDI is a condition specific or patient completed questionnaire comprising of 10 items to evaluate pain, and functional status which is mostly used for reporting neck pain. Each item on scale is scored from 0-5, where all the scores are added to total points and interpreted as percentages i.e. 0 point or 0% means no activity limitation and 50 points or 100% means complete activity limitation.

SECONDARY OUTCOMES:
Visual Analogue Scale | baseline and 2 weeks
  It is 10cm or 10nm line psychometric response scale to measure pain. Aggregate score ranges from 0-10. Score 0-4 means mild pain, 4-7 means moderate pain and 7- 10 means severe pain
Range of Motion | baseline and 2 weeks
  The universal goniometer (UG) is a measuring tool commonly used in clinics, to measure active cervical range of motion (ACROM), UG will be used to measure cervical ranges in all directions i.e. flexion, extension, lateral flexion and rotation. To measure cervical flexion and extension the UG axis will be placed over the external auditory meatus and will asked the patient will be asked to flex and extend the head, for lateral flexion over centre of sternal notch and for the cervical rotation over the centre of subject's head
WHO Quality of life-BREF (WHOQOL BREF) | baseline and 2 weeks
  The WHOQOL-BREF is an instrument which is used to assess psychometric properties. Consisting of 26 questions related to the following 4 domains: physical, psychological health, social relationship and environment. Each item is rated on 5-point scoring scale where each score is transferred between 0 and 100.

CONTACTS AND LOCATIONS:
Overall Officials: Zainab K Khan, MSAP, Principal Investigator — DUHS
Locations (1):
- Dow university of health sciences & Institute of physical medicine and rehabilitation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hurwitz EL, Randhawa K, Yu H, Cote P, Haldeman S. The Global Spine Care Initiative: a summary of the global burden of low back and neck pain studies. Eur Spine J. 2018 Sep;27(Suppl 6):796-801. doi: 10.1007/s00586-017-5432-9. Epub 2018 Feb 26. PMID 29480409
- [Background] de Campos TF, Maher CG, Steffens D, Fuller JT, Hancock MJ. Exercise programs may be effective in preventing a new episode of neck pain: a systematic review and meta-analysis. J Physiother. 2018 Jul;64(3):159-165. doi: 10.1016/j.jphys.2018.05.003. Epub 2018 Jun 19. PMID 29908853
- [Background] Rodriguez-Fuentes I, De Toro FJ, Rodriguez-Fuentes G, de Oliveira IM, Meijide-Failde R, Fuentes-Boquete IM. Myofascial Release Therapy in the Treatment of Occupational Mechanical Neck Pain: A Randomized Parallel Group Study. Am J Phys Med Rehabil. 2016 Jul;95(7):507-15. doi: 10.1097/PHM.0000000000000425. PMID 26745225
- [Background] Hoy D, March L, Woolf A, Blyth F, Brooks P, Smith E, Vos T, Barendregt J, Blore J, Murray C, Burstein R, Buchbinder R. The global burden of neck pain: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1309-15. doi: 10.1136/annrheumdis-2013-204431. Epub 2014 Jan 30. PMID 24482302
- [Background] Moradi-Lakeh M, Forouzanfar MH, Vollset SE, El Bcheraoui C, Daoud F, Afshin A, Charara R, Khalil I, Higashi H, Abd El Razek MM, Kiadaliri AA, Alam K, Akseer N, Al-Hamad N, Ali R, AlMazroa MA, Alomari MA, Al-Rabeeah AA, Alsharif U, Altirkawi KA, Atique S, Badawi A, Barrero LH, Basulaiman M, Bazargan-Hejazi S, Bedi N, Bensenor IM, Buchbinder R, Danawi H, Dharmaratne SD, Zannad F, Farvid MS, Fereshtehnejad SM, Farzadfar F, Fischer F, Gupta R, Hamadeh RR, Hamidi S, Horino M, Hoy DG, Hsairi M, Husseini A, Javanbakht M, Jonas JB, Kasaeian A, Khan EA, Khubchandani J, Knudsen AK, Kopec JA, Lunevicius R, Abd El Razek HM, Majeed A, Malekzadeh R, Mate K, Mehari A, Meltzer M, Memish ZA, Mirarefin M, Mohammed S, Naheed A, Obermeyer CM, Oh IH, Park EK, Peprah EK, Pourmalek F, Qorbani M, Rafay A, Rahimi-Movaghar V, Shiri R, Rahman SU, Rai RK, Rana SM, Sepanlou SG, Shaikh MA, Shiue I, Sibai AM, Silva DAS, Singh JA, Skogen JC, Terkawi AS, Ukwaja KN, Westerman R, Yonemoto N, Yoon SJ, Younis MZ, Zaidi Z, Zaki MES, Lim SS, Wang H, Vos T, Naghavi M, Lopez AD, Murray CJL, Mokdad AH. Burden of musculoskeletal disorders in the Eastern Mediterranean Region, 1990-2013: findings from the Global Burden of Disease Study 2013. Ann Rheum Dis. 2017 Aug;76(8):1365-1373. doi: 10.1136/annrheumdis-2016-210146. Epub 2017 Feb 16. PMID 28209629
- [Background] Kashyap R, Iqbal A, Alghadir AH. Controlled intervention to compare the efficacies of manual pressure release and the muscle energy technique for treating mechanical neck pain due to upper trapezius trigger points. J Pain Res. 2018 Dec 12;11:3151-3160. doi: 10.2147/JPR.S172711. eCollection 2018. PMID 30588067
- [Background] Cathcart E, McSweeney T, Johnston R, Young H, Edwards DJ. Immediate biomechanical, systemic, and interoceptive effects of myofascial release on the thoracic spine: A randomised controlled trial. J Bodyw Mov Ther. 2019 Jan;23(1):74-81. doi: 10.1016/j.jbmt.2018.10.006. Epub 2018 Oct 24. PMID 30691766
- [Background] Childs JD, Cleland JA, Elliott JM, Teyhen DS, Wainner RS, Whitman JM, Sopky BJ, Godges JJ, Flynn TW; American Physical Therapy Association. Neck pain: Clinical practice guidelines linked to the International Classification of Functioning, Disability, and Health from the Orthopedic Section of the American Physical Therapy Association. J Orthop Sports Phys Ther. 2008 Sep;38(9):A1-A34. doi: 10.2519/jospt.2008.0303. Epub 2008 Sep 1. PMID 18758050
- [Background] Thomas E, Cavallaro AR, Mani D, Bianco A, Palma A. The efficacy of muscle energy techniques in symptomatic and asymptomatic subjects: a systematic review. Chiropr Man Therap. 2019 Aug 27;27:35. doi: 10.1186/s12998-019-0258-7. eCollection 2019. PMID 31462989
- [Background] Rodriguez-Huguet M, Gil-Salu JL, Rodriguez-Huguet P, Cabrera-Afonso JR, Lomas-Vega R. Effects of Myofascial Release on Pressure Pain Thresholds in Patients With Neck Pain: A Single-Blind Randomized Controlled Trial. Am J Phys Med Rehabil. 2018 Jan;97(1):16-22. doi: 10.1097/PHM.0000000000000790. PMID 28678033
- [Background] Phadke A, Bedekar N, Shyam A, Sancheti P. Effect of muscle energy technique and static stretching on pain and functional disability in patients with mechanical neck pain: A randomized controlled trial. Hong Kong Physiother J. 2016 Apr 14;35:5-11. doi: 10.1016/j.hkpj.2015.12.002. eCollection 2016 Dec. PMID 30931028
- [Background] Louw S, Makwela S, Manas L, Meyer L, Terblanche D, Brink Y. Effectiveness of exercise in office workers with neck pain: A systematic review and meta-analysis. S Afr J Physiother. 2017 Nov 28;73(1):392. doi: 10.4102/sajp.v73i1.392. eCollection 2017. PMID 30135909
- [Derived] Khan ZK, Ahmed SI, Baig AAM, Farooqui WA. Effect of post-isometric relaxation versus myofascial release therapy on pain, functional disability, rom and qol in the management of non-specific neck pain: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Jun 13;23(1):567. doi: 10.1186/s12891-022-05516-1. PMID 35698187